CLINICAL TRIAL: NCT02967029
Title: Effect of Controlled Hypotension on Cerebral Oxygen Saturation in Patients Undergoing Functional Endoscopic Sinus Surgery: a Prospective Randomized Single Blind Clinical Trial
Brief Title: Effect of Controlled Hypotension on Cerebral Oxygen Saturation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Demet Altun, attending anesthesiologist, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IstanbulUn
Record Dates: First submitted 2016-11-07; First posted 2016-11-17 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Hypotension Drug-Induced; Cerebral Oxygen Saturation
MeSH Terms: conditions — Hypotension | interventions — esmolol; Remifentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- b group (Active Comparator): b group controlled hypotension with esmolol hydrochloride
  Interventions: Drug: Esmolol Hydrochloride
- r group (Active Comparator): r group controlled hypotension with remifentanil hydrochloride
  Interventions: Drug: Remifentanil Hydrochloride

INTERVENTIONS:
Drug: Esmolol Hydrochloride — the influence of brevibloc as a hypotensive agent on rSO2
  Other Names: Brevibloc 10 MG/ML Injectable Solution
  Arms: b group
Drug: Remifentanil Hydrochloride — the influence of remifentanyl as a hypotensive agent on rSO2
  Other Names: ultiva
  Arms: r group

SUMMARY:
For a successful functional endoscopic sinus surgery (FESS), it is crucial to provide effective controlled hypotension to reduce blood loss and provide a relatively blood-free surgical environment to facilitate surgery.

The goal of controlled hypotension is to maintain an arterial blood pressure which is sufficiently low to allow a reduction in bleeding with offering a superior intraoperative hemodynamic stability during stressful surgical events to maintain intact cerebral microcirculatory auto-regulation.

Auto-regulation impairment during controlled hypotension might increase oxygen extraction ratio. Thus monitoring the cerebral oxygen saturation (rSO2) to measure cerebral oxygenation becomes essential and it remains a challenge to clinically assess cerebral oxygenation on a routine basis.

Various recent studies reported based on facilitating the induction of controlled hypotension, but the effects of hypotension on cerebral perfusion and oxygenation and its effects on postoperative cognitive function are still poorly characterized. Moreover, the relationship between rSO2 and controlled hypotension has not been established in patients undergoing FESS.

Within the last decade, near infrared spectroscopy (NIRS) INVOS® monitors which is clinically most broadly spread technique, can be used for non-invasive assessment of cerebral perfusion by detecting changes in rSO2 by online monitoring of cerebral oxygenation.

In our clinical routine for achieving a controlled hypotension, esmolol and remifentanyl are the most commonly used hypotensive agents. The aim of this prospective randomized single blind study was to investigate the influence of remifentanyl as a hypotensive agent in comparison to esmolol on rSO2 by using NIRS and postoperative cognitive function in patients undergoing FESS.

DETAILED DESCRIPTION:
For a successful functional endoscopic sinus surgery (FESS), it is crucial to provide effective controlled hypotension to reduce blood loss and provide a relatively blood-free surgical environment to facilitate surgery.

The goal of controlled hypotension is to maintain an arterial blood pressure which is sufficiently low to allow a reduction in bleeding with offering a superior intraoperative hemodynamic stability during stressful surgical events to maintain intact cerebral microcirculatory auto-regulation.

Auto-regulation impairment during controlled hypotension might increase oxygen extraction ratio. Thus monitoring the cerebral oxygen saturation (rSO2) to measure cerebral oxygenation becomes essential and it remains a challenge to clinically assess cerebral oxygenation on a routine basis.

Various recent studies reported based on facilitating the induction of controlled hypotension, but the effects of hypotension on cerebral perfusion and oxygenation and its effects on postoperative cognitive function are still poorly characterized. Moreover, the relationship between rSO2 and controlled hypotension has not been established in patients undergoing FESS.

Within the last decade, near infrared spectroscopy (NIRS) monitors which is clinically most broadly spread technique, can be used for non-invasive assessment of cerebral perfusion by detecting changes in rSO2 by online monitoring of cerebral oxygenation.

In our clinical routine for achieving a controlled hypotension, esmolol and remifentanyl are the most commonly used hypotensive agents. The aim of this prospective randomized single blind study was to investigate the influence of remifentanyl as a hypotensive agent in comparison to esmolol on rSO2 by using NIRS and postoperative cognitive function in patients undergoing FESS.

After receiving the local institutional research ethics committee approval and written informed consent from each patient, 140 American Society of Anesthesiology (ASA) I and II patients aging between 18 and 65, undergoing for elective FESS and required controlled hypotension were enrolled in this study. Patients with hypertension, coronary artery diseases and cerebral insufficiency, severe hypovolemia and anemia, body mass index over 30 kg/m2, anticoagulation therapy and previous hypersensitivity to any of the study drugs were excluded from the study.

They were equally randomly assigned to receive either remifentanil or esmolol to maintain mean arterial blood pressure (MAP) between 55-65 mmHg.

After insertion of a peripheral venous cannula upon arrival to the operating room, balanced electrolyte solution at 5 ml/kg/h was initiated. Following the premedication with intravenous midazolam 0.05 miligram/kg IV 15 min prior to the induction of anesthesia, and standard monitoring was applied consisting of electrocardiography (EKG), noninvasive blood pressure, peripheral oxygen saturation (SPO2). Further, cerebral oxygen saturation value (rSO2, using the NIRS with adult probe placed in the median frontal region) was continuously monitored using NIRS before the induction of anesthesia.

After preoxygenation anaesthesia was induced with 2 miligram/kg propofol, 2 μg/kg fentanyl and to facilitate the endotracheal intubation 0.6 miligram/kg rocuronium was administered. Following orotracheal intubation, mechanical ventilation was adjusted to maintain PaCO2 at 35 to 40 mm Hg.

Anaesthesia maintenance was performed using sevoflurane (0.8 to 1 adjusted MAC) in a mixture of O2/Nitrous oxide 50%/50%. Then the treatment protocol consisting of remifentanil and esmolol were delivered in order to induce controlled hypotension that was considered effective when MAP reached the target pressure of 60 mmHg.

Patients in the esmolol group (Group E) received esmolol 0.5 miligram/kg iv at induction followed by a continuous infusion of esmolol 5-15 miligram/kg/min and titrated to the maximum dose 300μg/kg/min to reach target MAP of 50-60 mmHg about a value of 5 mmHg. Patients in the remifentanil group (Group R) received remifentanil 0.5 μg/kg/min at induction followed by an infusion of remifentanil 0.1- 0.5 μg/kg/min and titrated between 0,1- 0,5 μg/kg/min to reach target MAP of 50-60 mmHg about a value of 5 mmHg.

In both groups no surgical stress was applied during 5 min following start of hypotension.

Cerebral desaturation was defined as a reduction of rSO2 to higher than 20 % of baseline for ≥ 15 seconds. When cerebral desaturation occurred, remifentanil and esmolol infusion doses were decreased and MAP was increased with intravascular fluid administration and ephedrine. When hypotension below the target MAP and bradycardia below the heart rate 45 beats/min longer than one minute in duration were occurred, a bolus of ephedrine 10 mg iv and atropine 0.1 miligram/kg iv applied, respectively.

All operations were performed by the same attending surgeon in order to ensure consistency in the estimation of the surgical field who was blinded to the hypotensive agent. When MAP reached the desired range (50-60 mmHg) and was maintained for at least 10 minutes, the quality of the surgical field was defined in terms of blood loss and dryness using a 10 point scale (0= no bleeding, virtually bloodless field; 10= uncontrolled bleeding).

The cognitive function of the patients was assessed using Mini Mental State Examination (MMSE) test. Preoperative MMSE test was done at the premedication room 1 hour before surgery and 120 minutes after the discontinuation of the drugs for each patient. A decrease in the MMSE score ≥ 2 points from baseline was considered as an index of decline in cognitive function.

Hemodynamics (Diastolic blood pressure (DBP), Mean blood pressure (MBP), systolic blood pressure (SBP) and heart rate (HR), SPO2 and rSO2 were recorded preoperatively (baseline), postinduction 5th min (after administration of hypotensive and anesthetic agent), intraoperatively (10, 20, 30, 45, 60, 90 minutes), 5 and 10 minutes after stoppage of hypotensive agents. Additionally, the duration of surgery, duration of anesthesia, the consumption dose of hypotensive agents, desaturated and not desaturated patients among the groups were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) I and II patients
* aging between 18 and 65,
* undergoing for elective FESS
* requiring general anesthesia with endotracheal intubation

Exclusion Criteria:

* hypertension,
* coronary artery diseases and cerebral insufficiency,
* severe hypovolemia and anemia,
* body mass index over 30 kg/m2,
* anticoagulation therapy
* previous hypersensitivity to any of the study drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-11-01; Primary Completion 2017-07-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
cerebral desaturation | reduction of cerebral oxygen saturation to higher than 20 % of baseline for ≥ 15 seconds through surgery completion
  reduction of cerebral oxygen saturation to higher than 20 % of baseline for ≥ 15 seconds were recorded when MAP reached the desired range (50-60 mmHg)

SECONDARY OUTCOMES:
the quality of the surgical field | When MAP reached the desired range (50-60 mmHg) and was maintained for at least 10 minutes
  the quality of the surgical field was recorded in terms of blood loss and dryness using a 10 point scale (0= no bleeding, virtually bloodless field; 10= uncontrolled bleeding) When MAP reached the desired range (50-60 mmHg) and was maintained for at least 10 minutes
Arterial blood pressure | arterial blood pressure at baseline, after induction, peroperative and 5 and 10 minutes after stoppage of hypotensive agents through surgery completion
  Hemodynamic parameters as systolic, diastolic and mean arterial blood pressures were recorded preoperative, after induction, peroperative and 5 and 10 minutes after stoppage of hypotensive agents
Heart rate | Heart rate at baseline, after induction, peroperative and 5 and 10 minutes after stoppage of hypotensive agents through surgery completion
  Hemodynamic parameters as heart rates were recorded preoperative, after induction, peroperative and 5 and 10 minutes after stoppage of hypotensive agents
SPO2 value | SPO2 value at baseline, after induction, peroperative and 5 and 10 minutes after stoppage of hypotensive agents through surgery completion
  Hemodynamic parameters as SPO2 values were recorded preoperative, after induction, peroperative and 5 and 10 minutes after stoppage of hypotensive agents
cognitive function of the patients | cognitive function of the patients were assessed 1 hour before surgery and 120 minutes after the discontinuation of the drugs
  The cognitive function of the patients was assessed using Mini Mental State Examination (MMSE) test was recorded 1 hour before surgery and 120 minutes after the discontinuation of the drugs
the duration of surgery | duration of the surgery from the beginning of the surgery up to the end of the surgery
  duration of the surgery was recorded from the beginning of the surgery to the end of the surgery
duration of anesthesia | Intraoperative
  duration of anesthesia was recorded from the monitoring of the patient to the extubation of the patient
the consumption dose of hypotensive agents | Intraoperative
  the consumption dose of hypotensive agents were recorded from the from the beginning of the infusion to the stoppage of the drugs
desaturated and not desaturated patients among the groups | Intraoperative
  desaturated and not desaturated patients were recorded patients among the groups during the controlled hypotension
cerebral oxygen saturation | Intraoperative
  cerebral oxygen saturation was recorded when mean arterial pressure reached the target range (50-60 mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Demet Altun, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Department of Anesthesiology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No